CLINICAL TRIAL: NCT03970161
Title: Evaluation of Early Retinal Nerve Injury in Type 2 Diabetes Patients Without Diabetic Retinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiang Zhu, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Retinal nerve injury in T2DM
Record Dates: First submitted 2019-05-22; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Diabetic Retinopathy; Nerve Injury
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T2DM Patients (Experimental): Patients without microangioma changes undergoing FFA examination were included in the present study. All of the participants enrolled in the present study underwent a systematic ophthalmic examination.
  Interventions: Device: routine ophthalmic examination
- healthy control subjects (Experimental): All of the participants enrolled in the present study underwent a systematic ophthalmic examination.
  Interventions: Device: routine ophthalmic examination

INTERVENTIONS:
Device: routine ophthalmic examination — Routine ophthalmic examination, including slit lamp, intraocular pressure, and fundus examinations using direct or indirect ophthalmoscopy after pupil dilation and optical coherence tomography (OCT) examination. Patients with DM also underwent fundus fluorescein angiography (FFA) examination.

SUMMARY:
The object of this study is to investigate the damage to the retinal nerve fiber layer (RNFL) and ganglion cell complex layer (GCL+) in diabetic patients without retinal microangioma as detected by fundus fluorescein angiography (FFA) and to determine the kind of nerve damage more likely to indicate early injury.

DETAILED DESCRIPTION:
Patients with type 2 diabetes mellitus and healthy volunteers will be included in our study. Patients with retinal microangioma are excluded by FFA. The parameters around the optic disc and macular area of the above two groups are measured by optical coherence tomography (OCT), and the results will be analyzed using the SPSS 22.0 software.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM
2. Patients without microangioma

Exclusion Criteria:

1. Patients with any other ocular disease that might affect retinal nerve injury
2. Patients with optic neuropathy, age-related macular degeneration, retinal and choroidal disease, and retinal artery/vein occlusion.
3. Patients with hypertension, hematopathy, neuropathy, and other systemic diseases causing retinal nerve changes.
4. Patients with keratopathy, cataract, and vitreous hemorrhage were also excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2019-05-29 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Peripapillary RNFL thickness | 96 weeks
  Peripapillary RNFL thickness
GCL+ in the macular area obtained using the 3D wide mode | 96 weeks
  GCL+ in the macular area obtained using the 3D wide mode
Retinal thickness in all macular regions | 96 weeks
  Retinal thickness in all macular regions
RNFL thickness in the macular area obtained using the 3D Macula (v) mode | 96 weeks
  RNFL thickness in the macular area obtained using the 3D Macula (v) mode
GCL+ thickness in the macular region obtained using the 3D Macula (v) mode | 96 weeks
  GCL+ thickness in the macular region obtained using the 3D Macula (v) mode

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Zhu, Dorctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No